CLINICAL TRIAL: NCT02328235
Title: Effect of High Fat Diet on Muscle Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kevin Davy (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor-Investigator, Kevin Davy, Professor, Virginia Polytechnic Institute and State University
Organization: Virginia Polytechnic Institute and State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 06-367
Record Dates: First submitted 2014-12-22; First posted 2014-12-31 (Estimated); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Diabetes
Keywords: skeletal muscle, metabolism, physiology
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- High Saturated Fat Diet (Experimental): Subjects will receive a high fat diet for 5 day following a 2 week lead in diet. Measurements will be made pre-post high fat diet
  Interventions: Other: High Saturated Fat Diet

INTERVENTIONS:
Other: High Saturated Fat Diet — Prior to the high fat diet and after baseline testing, subjects will be asked to eat a standard diet to "lead-in" to the high fat diet condition. The diet will contain 55% of calories as carbohydrate, 30% as fat, and 15% as protein. The high fat diet will contain 50-60% of calories as fat, 20-30% as carbohydrate, and 10-20% as protein. Subjects will be provided with all of their meals throughout the study.

SUMMARY:
Skeletal muscle burns a significant amount of the fat and sugar that circulates in the blood stream. Ideally, when sugar is elevated in the blood stream, the muscle will either use it to make new energy or store it for later use. Likewise, for fatty acids. Skeletal muscle of obese and diabetic humans has been shown to inadequately use either sugar or fatty acids when they increase in the blood stream, and this has been termed metabolic inflexibility. The cause of metabolic inflexibility is not known, but it is believed that eating more fat than the body needs for energy may be a contributing factor. Metabolic inflexibility in skeletal muscle is bad because if the muscle does not use the sugar or fat, it will be stored elsewhere in the body and potentially lead to obesity and the resistance to insulin. The investigators have performed a research study with nonobese, healthy humans during which we fed them a high fat diet for 5 days. Interesting, only 5 days of a high fat diet is sufficient to cause the skeletal muscle to become metabolically inflexible just like that observed in obese and diabetic humans. The investigators are proposing addition studies to feed healthy humans a high fat diet for 5 days in effort to better understand what causes metabolic flexibility. The investigators are speculating that a high fat diet causes the intestines to release a substance called endotoxin that causes muscle to become metabolically inflexible. The investigators will test this notion in our proposed studies.

DETAILED DESCRIPTION:
Objective: To discern the potential mechanism(s) by which high saturated fat feeding disrupts normal skeletal muscle metabolism. Our working hypothesis is that high saturated fat feeding increases gut permeability and blood endotoxin, which elicits pro-inflammatory signaling in skeletal muscle and alters the normal adaptive response to a meal. Preliminary evidence using a model of acute (5 days), high saturated fat feeding, isocaloric to habitual intake, in healthy, non-obese humans is presented herein to support this hypothesis.

Background: The inability for skeletal muscle to adapt fuel oxidation to fuel availability is termed metabolic inflexibility, a well characterized feature of disease states such as obesity, metabolic syndrome, and type 2 diabetes (T2D). The mechanism(s) responsible for skeletal muscle metabolic inflexibility are not known. Recently, there has been growing interest in the role of gut permeability and blood endotoxin in the pathology of metabolic derangements associated with obesity and T2D. Rodent studies have revealed direct links between the gut microbiome and metabolic disease, as well as associations between elevated blood endotoxin and metabolic dysregulation, both at the whole body and tissue level. High fat feeding in rodents is known to elicit elevated levels of blood endotoxin, a phenomenon that is termed metabolic endotoxemia. In humans, obesity and T2D are associated with increased blood endotoxin and single meals have been shown to elevate blood endotoxin, but to date, there is no evidence in humans that high fat feeding results in metabolic endotoxemia. Moreover, there are no established links between gut permeability, metabolic endotoxemia, and skeletal muscle metabolic function in humans.

Approach. We are proposing to utilize a model of acute high fat feeding in healthy humans to study the interplay between gut function, blood endotoxin, and skeletal muscle pro-inflammatory signaling and metabolic adaptability. We will employ a two-week lead-in period, during which research participants will be fed prepared meals that are isocaloric to their habitual diet, followed by five days of high saturated fat feeding. The high saturated fat feeding period will consist of prepared meals that are isocaloric to habitual diet with a macronutrient composition of 50% fat (45% of which will be saturated fat), 35% carbohydrate, and 15% protein. Studying healthy, nonobese humans in this context is an innovative approach on two levels: 1) any confounding influences associated with metabolic disease (obesity, diabetes, or metabolic syndrome) are eliminated, e.g., insulin resistance, hyperlipidemia, impaired gut function, pre-existing metabolic dysfunction and inflammatory tone; and 2) the isocaloric feeding design negates the confounding influence of a positive energy balance and allows us to specifically examine the effects of acutely increasing dietary saturated fat.

ELIGIBILITY:
Inclusion Criteria:

* Males, age 18-40 years; BMI between 20 and 30 kg/m2. Weight stable for previous 6 months (± 2.0kg).

Sedentary to recreationally active (≤ 3 days, 20 min/day of walking type exercise, no planned exercise other than leisure walking for transportation purposes).

Verbal and written informed consent

non-smoking

Approved for participation by Medical Director (Jose Rivero, M.D.)

Exclusion Criteria:

* 1. Past or current ischemic heart disease, stroke, respiratory disease, endocrine or metabolic disease, neurological disease, or hematological-oncological disease

  2. Family history of diabetes

  3. BMI > 30 kg/m2, blood pressure > 140/90 mmHg or antihypertensive medications, fasting glucose > 100 mg/dl, LDL cholesterol > 130 mg/dl, total cholesterol > 200 mg/dl, triglycerides > 250 mg/dl.

  4. Verbal and written informed consent

  4. Smoking, alcohol consumption > 2 servings/d, or taking medications (including but not limited to statins or other drugs with anti-inflammatory actions) or antioxidant vitamins or supplements, or know to affect carbohydrate or lipid metabolism.

  5. Total daily dietary fat consumption ≥ 35% and/or saturated fat consumption of ≥ 15%.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-03-09 (Actual)

PRIMARY OUTCOMES:
Metabolic Flexibility measured ex vivo in skeletal muscle using radio labeled carbon isotopes | 1 day
  Assess substrate handling ex vivo in skeletal muscle using radio labeled isotopes pre and post high fat diet

SECONDARY OUTCOMES:
Intestinal Permeability using a 4 sugar probe test and mass spectrometry | 24 hours
  Assess intestinal permeability with a variety of insoluble sugars and their level of excretion in the urine with mass spectrometry pre and post high fat diet

CONTACTS AND LOCATIONS:
Overall Officials: Kevin P Davy, PhD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Virginia Polytechnic and State University, Blacksburg, Virginia, United States